CLINICAL TRIAL: NCT04654650
Title: Prospective Registry and Biobank for Long-term Observational Studies in Adult Patients with Pulmonary Hypertension
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: HHPHBiobank
Record Dates: First submitted 2020-11-04; First posted 2020-12-04 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective registry and biobank for long-term observational studies in adult patients with pulmonary hypertension

DETAILED DESCRIPTION:
In a prospective registry prevalent and incident patients diagnosed with group 1 to 5 pulmonary hypertension will be enrolled. In an integrated biobank body fluid samples will be collected at enrollment and sequentially during treatment with targeted drugs for pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulmonary hypertension group 1 to 5
* Ability to give informed consent

Exclusion Criteria:

- Withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pulmonary hypertension and patients referred to a pulmonary hypertension center for suspected pulmonary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2041-01-25 (Estimated); Study Completion 2041-01-25 (Estimated)

PRIMARY OUTCOMES:
Transplant-free survival | Up to 20 years of follow-up after enrollment

SECONDARY OUTCOMES:
Risk score (averaging low, intermediate and high risk categories) as proposed by the 2015 European Society of Cardiology (ESC)/European Respiratory Society (ERS) guidelines for pulmonary hypertension | Up to 20 years of follow-up after enrollment
Registry to Evaluate Early And Long-term PAH Disease Management (REVEAL) 2.0 risk score | Up to 20 years of follow-up after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg, Germany